CLINICAL TRIAL: NCT03764488
Title: A Phase 1, Safety, Tolerability, and Distribution Study of a Microdose of Radiolabeled BIIB067 Co-administered With BIIB067 to Healthy Adults
Brief Title: A Study to Evaluate Safety, Tolerability, and Distribution of a Microdose of Radiolabeled BIIB067 (99mTc-MAG3-BIIB067) Co-administered With BIIB067 (Tofersen) to Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 233HV101
Record Dates: First submitted 2018-12-03; First posted 2018-12-05 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — tofersen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BIIB067 High Dose + 99mTc-MAG3-BIIB067 in 15 mL aCSF (Experimental): Participants will receive intrathecal injection consisting of unlabeled BIIB067 and 99mTc-MAG3-BIIB067 in 15 milliliter (mL) artificial cerebrospinal fluid (aCSF).
  Interventions: Drug: Tofersen; Drug: 99mTc-MAG3-BIIB067
- BIIB067 Low Dose + 99mTc-MAG3-BIIB067 in 15 mL aCSF (Experimental): Participants will receive intrathecal injection consisting of unlabeled BIIB067 and 99mTc-MAG3-BIIB067 in 15 mL aCSF.
  Interventions: Drug: Tofersen; Drug: 99mTc-MAG3-BIIB067
- BIIB067 Low Dose + 99mTc-MAG3-BIIB067 in 5 mL aCSF (Experimental): Participants will receive intrathecal injection consisting of unlabeled BIIB067 and 99mTc-MAG3-BIIB067 in 5 mL aCSF.
  Interventions: Drug: Tofersen; Drug: 99mTc-MAG3-BIIB067
- BIIB067 Low Dose + 99mTc-MAG3-BIIB067 in up to 20 mL aCSF (Experimental): Participants will receive intrathecal injection consisting of unlabeled BIIB067 and 99mTc-MAG3-BIIB067 in up to 20 mL aCSF.
  Interventions: Drug: Tofersen; Drug: 99mTc-MAG3-BIIB067

INTERVENTIONS:
Drug: Tofersen — Administered as specified in the treatment arm.
  Other Names: BIIB067; QALSODY
Drug: 99mTc-MAG3-BIIB067 — Administered as specified in the treatment arm.

SUMMARY:
The primary objective of the study is to evaluate the distribution in the central nervous system (CNS) of a microdose 99mTc-MAG3-BIIB067 co-administered with unlabeled BIIB067 (Tofersen). The secondary objective of the study is to assess the safety and tolerability of unlabeled BIIB067 co-administered with a microdose of 99mTc-MAG3-BIIB067 to healthy participants.

ELIGIBILITY:
Key Inclusion Criteria:

* Must have a body mass index between 18 and 30 kilogram per square meter (kg/m^2), inclusive.
* All men must practice highly effective contraception during the study and for 5 months after their last dose of study treatment.
* All female participants must be of non-childbearing potential and must meet 1 of the following criteria to participate in the study: a. Postmenopausal, b. History of bilateral oophorectomy (performed at least 6 weeks prior to Screening), c. History of hysterectomy (performed at least 6 weeks prior to Screening), or d. History of female surgical sterilization (e.g., bilateral tubal ligation; performed at least 6 weeks prior to Screening).

Key Exclusion Criteria:

* History of or ongoing clinically significant cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, or other major disease, as determined by the Investigator.
* Clinically significant abnormal laboratory test values, as determined by the Investigator, at Screening or Check-in.
* Use of any prescription medication, over-the-counter medication (e.g., aspirin and nonsteroidal anti-inflammatory drugs [excluding acetaminophen]), or dietary and herbal supplements (e.g., St. John's wort) within 28 days of Check-in and an unwillingness to refrain from use through end of study (i.e., through the Day 91 visit), unless specifically permitted elsewhere within the protocol.
* Current enrollment in any other drug, biologic, device, or clinical study, or treatment with an investigational drug or approved therapy for investigational use within 30 days (6 months for biologics) or 5 half-lives, whichever is longer, prior to Check-in.
* History or physical examination that could be suggestive of a medical or mechanical condition, disorder, or disease that could represent a relative contraindication to lumbar puncture (LP), including but not limited to: (a) medication use that prolongs coagulation times, including aspirin; (b) known disorders of the coagulation cascade, platelet function, or platelet count; (c) low white blood cell counts; (d) chronic low back pain; (e) prior lumbar spine surgery; (f) anatomical factors at or near the LP site; (g) clinical signs of raised intracranial pressure (e.g., headache, papilledema, or focal neurologic signs).
* Contraindications to radiation exposure for research purposes.
* Exposure to ionizing radiation within the last 12 months that would result in approaching the exposure limits for healthy volunteers.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2021-07-10 (Actual)

PRIMARY OUTCOMES:
BIIB067 Concentrations Throughout the CNS | 1 to 24 hours post-dose on Day 1
  BIIB067 concentrations throughout the CNS will be estimated by single-photon emission computed tomography (SPECT)/computed tomography (CT) imaging of 99mTc-MAG3-BIIB067.

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to Day 91
  An AE is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An SAE is any untoward medical occurrence that at any dose: results in death, in the view of the Investigator, places the participant at immediate risk of death (a life-threatening event), however, this does not include an event that, had it occurred in a more severe form, might have caused death; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; results in a congenital anomaly/birth defect or is a medically important event.
Dose of Radiation Absorbed (Dosimetry) in Specific Regions of the CNS | 1 to 24 hours post-dose on Day 1
  Dose of radiation absorbed (dosimetry) in specific regions of the CNS will be estimated by SPECT/CT imaging of 99mTc-MAG3-BIIB067.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (2):
- United States (2):
  - Research Site, Boston, Massachusetts
  - Research Site, New York, New York